CLINICAL TRIAL: NCT06066268
Title: Role of microRNAs in Critical Limb Ischemia
Brief Title: miRNAs in Critical Limb Ischemia (miRNACLI)
Acronym: miRNACLI
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Fabio Martelli, Dr., IRCCS Policlinico S. Donato
Other Study IDs: miRNACLI
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Critical Limb Ischemia
Keywords: microRNA; Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — muscle biopsis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1) Critical limb ischemia (CLI);: 1)Critical limb ischemia (CLI):
  * Patients suffering from CLI undergoing lower limb revascularization via subgenual femoropopliteal bypass. muscle biopsies willbe taken.
  * Patients suffering from terminal CLI and/or gangrene of the lower limb undergoing thigh amputation. Muscle biopsies will be taken.
  * Patients suffering from terminal CLI and/or gangrene of the lower limb undergoing leg amputation. Muscle biopsies will be taken.
  Interventions: Diagnostic Test: Critical limb ischemia: analysis of RNAs
- 2)Controls: 2)Controls: patients affected by infrarenal abdominal aortic aneurysm (AAA) free from CLI, affected and not affected by type 2 diabetes mellitus, undergoing endovascular exclusion surgery of the AAA (EVAR), similar by age and sex to CLI patients. Sartorius muscle biopsies will be taken.
  Interventions: Diagnostic Test: Controls: analysis of RNAs

INTERVENTIONS:
Diagnostic Test: Critical limb ischemia: analysis of RNAs — analysis of miRNA expression levels
  Groups: 1) Critical limb ischemia (CLI);
Diagnostic Test: Controls: analysis of RNAs — analysis of miRNAs expression levels
  Groups: 2)Controls

SUMMARY:
For the present study, 40 patients affected by critical limb ischemia of different severity will be enrolled: patients affected by critical limb ischemia undergoing subgenual femoropopliteal bypass; patients suffering from terminal ischemia causing gangrene and therefore undergoing major amputation of the lower limb. Biopsies from the first 20 enrolled patients will be used for miRNA profiling. The total of 40 biopsies obtained from all enrolled patients will instead be used for the validation of the miRNAs identified in the profiling.

The results obtained will be compared with those obtained in 40 control patients affected by infrarenal abdominal aortic aneurysm (AAA) undergoing endovascular exclusion surgery (EVAR) of the AAA without any ischemia of the lower limbs. Also in this case the biopsies of the first 20 control patients enrolled will be used for miRNA profiling. The total of 40 biopsies obtained from all control patients will instead be used for the validation of the miRNAs identified in the profiling. A total of 80 patients (40 cases and 40 controls) will be enrolled.

DETAILED DESCRIPTION:
The analyzes of the expression of miRNAs and the RISC complex will be carried out on fragments of skeletal muscle taken from different sites depending on whether they are cases or controls.

Cases:

* Patients suffering from CLI undergoing lower limb revascularization via subgenual femoropopliteal bypass: Gastrocnemius muscle biopsies will be taken.
* Patients suffering from terminal CLI and/or gangrene of the lower limb undergoing thigh amputation: biopsies will be taken in different muscle districts. In particular, biopsies of the Sartorius or Vastus lateralis muscle will be taken at the amputation site, both from the proximal muscle belly which remains covering the bone stump, and from the part of the muscle belly sacrificed with the amputated limb. Biopsies of the Gastrocnemius and Tibialis anterior muscles will be taken from the amputated leg.
* Patients suffering from terminal CLI and/or gangrene of the lower limb undergoing leg amputation: biopsies will be taken in different muscle districts. In particular, biopsies of the Gastrocnemius and Tibialis anterior muscles will be carried out at the amputation site, both from the proximal muscle belly which remains covering the bone stump, and from the part of the muscle belly sacrificed with the amputated limb.

Controls:

• The control subjects will be represented by individuals affected by infrarenal abdominal aortic aneurysm (AAA) free from CLI, affected and not affected by type 2 diabetes mellitus, undergoing endovascular exclusion surgery of the AAA (EVAR), similar by age and sex to CLI patients. Sartorius muscle biopsies will be taken.

The analyzes of the expression of circulating miRNAs will be carried out on 2 7 ml tubes of peripheral venous blood, taken before the surgical incision from the same cases and controls described in the previous point.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* patients affected by CLI candidates for popliteal exploration surgery and/or subgenual femoropopliteal bypass.
* Patients affected by CLI with irreversible ischemia and/or distal gangrene of the lower limb candidates for major amputation of the lower limb.

Controls:

• patients affected by infrarenal abdominal aortic aneurysm (AAA) undergoing endovascular exclusion surgery of the AAA (EVAR) who are free from CLI, affected and not affected by type 2 diabetes mellitus.

Exclusion Criteria:

* Pregnant women
* Patients carriers of genetic diseases
* Patients suffering from malignant neoplasia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical limb ischemia patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Identification of potentially pathogenic miRNAs in CLI and related target mRNAs. | 1 year to 10 years
  Identify miRNAs and their targets that directly interact with the RNA Induced Silencing Complex (RISC) in muscle biopsies obtained from CLI patients.
Identification of disease biomarkers | 1 year to 10 years
  Identify plasma miRNAs to be used as disease biomarkers that can be used to assess disease status and severity with a minimally invasive procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Martelli, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, Milan, Italy